CLINICAL TRIAL: NCT04027127
Title: The Effect of Serum Netrin-1 Levels on Diagnosis and Prognosis in Patients Presenting to the Emergency Department With Acute Coronary Syndrome
Brief Title: The Role of Netrin -1 in Acute Coronary Syndrome
Acronym: ACS-NETRİN-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, huseyin mutlu, Asst. Prof. Dr. Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: aksaray 2013-23
Record Dates: First submitted 2019-06-18; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome
Keywords: netrin-1; acs; reperfuzion
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: PATIENT AND CONTROL GROUP will be divided into two.
Who Masked: Participant
Masking Description: Patient group; Those diagnosed with ACS over 18 years of age, planned angiography and accepted angiography. The control group consisted of volunteers without disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACS GRUP (Active Comparator): Demographic characteristics, history, vital signs, laboratory findings, coronary angiography (CAG) and echocardiography (ECO) findings of the patients were recorded. Netrin-1 levels were studied with blood collected at the hospital and 6-8 hours after CAG. CAG results were evaluated by TIMI flow. The patients were divided into two groups with and without TIMI 3 flow and Netrin-1 levels were compared.
  GRACE (Global Registry of Acute Coronary Events) and TIMI (Thrombolysis in Myocardial Ischemia) clinical risk assessments were performed and Netrin-1 values were compared.
  Interventions: Other: netrin-1 value on admission to hospital
- plasebo grup (Active Comparator): It consisted of those without any disease and netri-1 values at admission were compared with the uptake patient group.
  Interventions: Other: netrin-1 value on admission to hospital

INTERVENTIONS:
Other: netrin-1 value on admission to hospital

SUMMARY:
In our study, Netrin -1; We found that patients with ACS increased at the time of admission, decreased TIMI 3 flow after angiography, and higher risk groups in high risk groups such as TIMI and GRACE were found to have higher Netrin-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* diagnose ACS
* patients undergoing angiography

Exclusion Criteria:

* CVE history
* Neurological disease
* Pregnancy and Lactation
* Liver failure
* Diagnosed malignity
* Use of anticonvulsant and nephrotoxic medication
* Chronic kidney disease
* Not having angiography
* Developing acute renal failure after angiography
* Patients who rejected to participate were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-09-15 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
serum netrin-1 value | 30 minute
  Netrin-1 in plasma was measured by enzyme-linked immunosorbent assay (ELISA) (Mybıosource MBS044526 ) All assays were performed in duplicate. Plasma Netrin-1 is expressed in picograms (pg) per mg.

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Mutlu, MD, Study Director — Aksaray/Turkey

IPD SHARING:
Plan to Share IPD: No